CLINICAL TRIAL: NCT02347358
Title: Mechanical Opening Device Implantation Following Intravenous r-tPA and Recanalization Outcome Evaluation in Stroke Disease (MODIFIED) Trial
Brief Title: Mechanical Opening Device Implantation Following Intravenous r-tPA for Recanalization in Acute Ischemic Stroke
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Artillery General Hospital (Other)
Collaborators: Hunan Rui Kang Tong technology development co., LTD (Unknown)
Responsible Party: Principal Investigator, Weijian Jiang, Principal Investigator, The Second Artillery General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013CB733805
Record Dates: First submitted 2015-01-10; First posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Ischemic Cerebrovascular Accident
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV r-tPA with JRecanTM blood FR device (Experimental): Dual IV r-tPA therapy and adjunctive treatment with JRecanTM blood flow recanalisation device
  Interventions: Device: JRecanTM blood FR device
- IV r-tPA (Active Comparator): IV infusion of r-tPA
  Interventions: Drug: IV r-tPA

INTERVENTIONS:
Device: JRecanTM blood FR device — JRecanTM blood flow recanalisation device
  Arms: IV r-tPA with JRecanTM blood FR device
Drug: IV r-tPA — intravenous recombinant human tissue plasminogen activator
  Other Names: intravenous recombinant human tissue plasminogen activator
  Arms: IV r-tPA

SUMMARY:
This study is to test a hypothesis that temporary implantation of JRecanTM blood flow recanalisation device within 6.5 hours of symptom onset of acute ischemic stroke due to a major intracranial artery occlusion following IV r-tPA can provide a greater rate of early successful recanalisation than treatment of IV r-tPA alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75
2. Clinical presentations consistent with acute ischemic stroke
3. NIHSS ≥ 8 and < 30 at the time of randomization
4. Initiation of the correct IV t-PA dose treatment within 4.5 hours of onset of stroke symptoms (onset time is defined as the last time when the patient was witnessed to be at baseline)
5. Complement of catheter angiography within 6.5 hours of onset of stroke symptoms
6. Thrombolysis in myocardial Infarction (TIMI) 0-1 flow in the intracranial internal carotid artery, M1 segment of the MCA, basilar artery, or intracranial vertebral artery with contralaterally chronic intracranial vertebral artery occlusion confirmed by catheter angiography
7. The acute occlusion lesion is accessible to the JRecanTM blood flow recanalisation device
8. Functional independence before this time stroke (Modified Rankin Score ≤ 1)
9. Subject or subject's legally authorized representative has signed and dated an Informed Consent Form according to country regulations, ethics committee requirements.
10. Subject is willing to conduct protocol-required follow-up visits.

Exclusion Criteria:

1. NIHSS <8 or ≥30
2. Rapid neurological improvement prior to study randomization
3. Female who is pregnant or lactating or has a positive pregnancy test at time of admission
4. Taking part in another clinical study.
5. History of stroke in the past 3 months.
6. Current participation in another investigational drug or device treatment study.
7. Uncontrolled hypertension defined as systolic blood pressure > 185 or diastolic blood pressure > 110 that cannot be controlled except with continuous parenteral antihypertensive medication.
8. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency. (Patients without history or suspicion of coagulopathy do not require INR or prothrombin time lab results to be available prior to enrollment.)
9. Warfarin therapy with INR greater than 1.7.
10. Low molecular Weight Heparins (such as Dalteparin, Enoxaparin, Tinzaparin, Fondaparinux) as DVT prophylaxis or in full dose within the last 24 hours from screening.
11. Subject who has received heparin or a direct thrombin inhibitor (e.g. rivaroxaban, Angiomax™, argatroban, Refludan™) within the last 48 hours must have a normal partial thromboplastin time (PTT) to be eligible.
12. Subject who has received factor Xa inhibitor therapy (e.g. dabigatran) within the past 24 hours must have a normal ecarin clotting time to be eligible. Subject who has received factor Xa inhibitor therapy more than 24 hours ago but less than 48 hours ago must have a normal partial thromboplastin time (PTT) to be eligible.
13. Baseline lab values: glucose < 50 mg/dl or > 400 mg/dl, platelets < 100,000, or Hct < 25.
14. Renal Failure as defined by a serum creatinine > 2.0 or Glomerular Filtration Rate [GFR] < 30.
15. Subject who requires hemodialysis or peritoneal dialysis, or who have a contraindication to an angiogram for whatever reason.
16. Life expectancy of less than 90 days.
17. Previous intra-cranial hemorrhage, neoplasm, subarachnoid hemorrhage, cerebral aneurysm, or arteriovenous malformation.
18. Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal.
19. Presumed septic embolus, or suspicion of bacterial endocarditis.
20. Presumed pericarditis including pericarditis after acute myocardial infarction.
21. Suspicion of aortic dissection.
22. Surgery or biopsy of parenchymal organ within 30 days.
23. Trauma with internal injuries or ulcerative wounds within 30 days.
24. Severe head trauma or head trauma with loss of consciousness within 90 days.
25. Any active or recent hemorrhage within 30 days.
26. Cerebral vasculitis.
27. Subject with a pre-existing neurological or psychiatric disease that would confound the neurological and functional evaluations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Early successful recanalisation (assessed by the imaging core laboratory) | 24 hours
  TIMI（thrombolysis in myocardial infarction）2 or 3 recanalisation 1 hour after enrollment blindly assessed by the imaging core laboratory and without any presence of symptomatic intracranial hemorrhage within 24 hours blindly assessed by independent neurologists.

SECONDARY OUTCOMES:
Good neurological outcome( modified Rankin Scale (mRS) score ≤2, or National Institutes of Health Stroke Scale（NIHSS）score improvement of 10 points or more) | 90 days
  modified Rankin Scale (mRS) score ≤2, or National Institutes of Health Stroke Scale（NIHSS）score improvement of 10 points or more.
Incidence of device related and procedure-related serious adverse events(SAEs) | 30 days
  The incidence of device related and procedure-related serious adverse events(SAEs)
Additional safety end-points (symptomatic intracranial haemorrhage at 24 hours, and Death due to any cause at 90 days) | 90 days
  symptomatic intracranial haemorrhage at 24 hours, and Death due to any cause at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Jiang, MD,PhD, Principal Investigator — New Era Stroke Care and Research Institute, The Second Artillery General Hospital Beijing